CLINICAL TRIAL: NCT02309307
Title: A Prospective, Open Label, Single Arm, Multi-center Study to Assess the Safety and Performance of a Soft Tissue Repair Device (VergenixTM STR) in Patients With Epicondylitis (Tennis Elbow)
Brief Title: Tissue Repair Device (VergenixTM STR) in Patients With Epicondylitis (Tennis Elbow)
Acronym: CP-STR-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Collplant (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-STR-01
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2015-01

CONDITIONS: Non Ruptured Tendon Injuries; Tendinopathy
Keywords: safety and performance
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 Tissue Repair Device (Experimental): Tissue Repair Device
  Interventions: Device: Tissue Repair Device (VergenixTM STR)

INTERVENTIONS:
Device: Tissue Repair Device (VergenixTM STR) — Administration of Soft Tissue Repair Device

SUMMARY:
The VergenixTM STR device is intended for the repair of non ruptured tendon injuries (Tendinopathy).

DETAILED DESCRIPTION:
The VergenixTM STR device is an advanced Soft tissue repair device, made of lyophilized Type I rhCollagen and Calcium Chloride that will be mixed with autologous PRP prior to injection for the repair of non ruptured tendon injuries (Tendinopathy). Three (3) ml of the mixed solution will be injected into the common extensor tendon.

ELIGIBILITY:
Inclusion Criteria:

1. Man or woman aged 18 - 80 years old.
2. Clinical diagnosis of lateral epicondylitis based on site of pain, pain

   elicited with active extension of the wrist in pronation and elbow

   extension.
3. Documented ultrasonography diagnosis of common extensor

   tendinosis and possible tear based on abnormal echotexture (tendon

   thickening, anechoic areas, areas of hypoechogencicity, loss of

   fibrillar pattern).
4. Chronic symptoms (equal or greater than 3 months).
5. PRTEE questionnaire score of at least 50 out of 100.
6. For child-bearing potential females, documentation of birth

   control.
7. Signing informed consent form. -

Exclusion Criteria:

1. Acute symptom onset (less than 3 months).
2. History of acute elbow trauma.
3. History of Rheumatoid Arthritis.
4. History of Inflammatory disease
5. History of Fibromyalgia
6. The patient has active malignant disease of any kind. A patient who

   has had a malignant disease in the past, was treated and is currently

   disease-free for at least 5 years, may be considered for study entry.
7. The patient is treated with anti-coagulant medication
8. The patient previously underwent a surgery for lateral

   epicondylitis.
9. The patient previously received local injections, including steroids

   within the last 30 days
10. Signs of other causes for lateral elbow pain (posterior interosseous

    nerve entrapment, osteochondral lesion).
11. Wounds around the elbow
12. Likely problems, in the judgment of the investigator, with maintaining follow-up.
13. Clinically significant abnormalities in hematology and blood

    chemistry lab tests at screening that in the opinion of the

    investigator might interfere with the patient's safety or participation

    in the study.
14. Known as positive HIV, hepatitis B, or hepatitis C.
15. Known history of a significant medical disorder, which in the

    investigator's judgment contraindicates the patient's participation.
16. Known hypersensitivity and/or allergy to collagen.
17. Drug or alcohol abuse (by history).
18. Pregnancy of child-bearing potential females.
19. Participation in another study within 30 days prior to screening

visit.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01-11 (Actual); Primary Completion 2016-08-24 (Actual); Study Completion 2016-08-24 (Actual)

PRIMARY OUTCOMES:
Changes in pain as a continuous outcome measure using the Patient-Rated Tennis Elbow Evaluation (PRTEE) questionnaire. | Up to 194 days
Functional Disability using the PRTEE questionnaire. | Up to 194 days
Tendon thickness (i.e tendon healing/improvement) and Doppler activity using US at 3M. | Up to 194 days
Health related Quality of life parameters questionnaire. | Up to 194 days
Pain free/maximum grip strength (Dynamometer) | Up to 194 days

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Hadassah MC, Jerusalem
  - Meir MC, Kfar Saba
  - Assaf Harofeh MC, Zrifin